CLINICAL TRIAL: NCT00405262
Title: The Effectiveness of Bupivicaine Infusion Versus Intravenous Ketorolac for Postoperative Analgesia After Iliac Crest Bone Harvesting for Lefort I Osteotomy or Alveolar Cleft Repair.
Brief Title: A Comparison of Bupivacaine and Ketorolac for Postoperative Analgesia After Iliac Crest Bone Harvesting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000008719
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Pain
Keywords: Pediatrics; Postoperative Analgesia; orthopedic surgery; Iliac Crest Bone Graft; Osteotomy; cleft palate
MeSH Terms: conditions — Pain, Postoperative; Cleft Palate | interventions — Ketorolac; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Ketorolac
- 2 (Experimental)
  Interventions: Drug: Bupivacaine
- 3 (Experimental)
  Interventions: Drug: ketorolac + bupivacaine

INTERVENTIONS:
Drug: Ketorolac — 0.5 mg•kg-1 IV at the end of surgery before extubation and then 3 additional doses every 8 hours thereafter
  Arms: 1
Drug: Bupivacaine — 0.2 mL•kg-1 (lean body mass) bolus of bupivacaine 0.25% with epinephrine 1:200 000 will be injected through the IC catheter at the end surgery before the patient's trachea is extubated to detect intravascular injection. An infusion of the same solution will be started at 0.1 mL•kg-1•hour-1 (lean body mass) for 24 hours.
  Arms: 2
Drug: ketorolac + bupivacaine — 0.2 mL•kg-1 (lean body mass) bolus of bupivacaine 0.25% with epinephrine 1:200 000 will be injected through the IC catheter at the end surgery before the patient's trachea is extubated to detect intravascular injection. An infusion of the same solution will be started at 0.1 mL•kg-1•hour-1 (lean body mass) for 24 hours.
  For ketorolac, patients will receive 0.5 mg•kg-1 IV at the end of surgery before extubation and then 3 additional doses every 8 hours thereafter
  Arms: 3

SUMMARY:
The efficacy of three postoperative pain management regimens will be compared in patients undergoing Lefort I osteotomy or alveolar cleft repair with Iliac crest bone grafts (ICBG) to determine the best way of managing postoperative pain.

DETAILED DESCRIPTION:
Iliac crest bone grafts (ICBG) are used for many types of surgeries including alveolar cleft repair, Lefort I osteotomies, spinal fusion, and fracture management. ICBG donor sites are notoriously painful, and the pain is often more severe than that from the primary operative site.

Postoperative pain management after operations that involve harvesting ICBG usually includes opioids, which are most often delivered by a patient-controlled device. Additional analgesics may include acetaminophen, non-steroidal anti-inflammatory (NSAID) drugs, and local anesthetic agents, such as bupivacaine or ropivacaine. Local anesthetics may also be injected intermittently or continuously into the wound via an indwelling catheter inserted at the time of surgery. All but one of these studies have shown a significant reduction in pain scores and opioid consumption using local anesthetic through an indwelling catheter.

Only one study has investigated the effects of NSAIDs on postoperative ICBG pain. This study found that intravenous ketorolac did not reduce morphine consumption. However, there was a trend to lower morphine use with ketorolac, and pain and patient satisfaction scores were not measured.

Currently, we do not use local anesthetic infusions via an indwelling iliac crest catheter for patients at our institution undergoing Lefort I osteotomy or alveolar cleft repair with ICBG since we find the above pain management regimen to be effective, with most patients using low to moderate amounts of morphine. To our knowledge, no study to date has compared the efficacy of ketorolac to local anesthetic infusions for patients undergoing Lefort I osteotomy or alveolar cleft repair with ICBG.

ELIGIBILITY:
Inclusion Criteria:

* Alveolar bone graft patients age 10-13 years of age
* Lefort I osteotomy patients needing ICBG age 14 to 20 years
* able to operate a patient-controlled analgesia (PCA) device

Exclusion Criteria:

* Allergy, sensitivity or contraindication to any non-steroidal anti-inflammatory drugs
* Allergy, sensitivity or contraindication to morphine
* History of gastric ulcer or bleeding diathesis

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain, assessed with a numerical analog system | As soon as the patient is able to respond appropriately and then approximately every 4 hours for 48 hours
Patient satisfaction score | 24 hours

SECONDARY OUTCOMES:
Morphine consumption | Every 4 hours
Total number of episodes of nausea, vomiting, and pruritis | 48 hours
Doses of all anti-emetics | 48 hours
Heart rate and respiratory rate variables | 48 hours
Time to first ambulation | Time determined by outcome
Wound healing at iliac crest site | 1, 4, 8 and 16 weeks post-operatively
X-ray data on recipient site | 1, 4, 8 and 16 weeks post-operatively
Clinical assessment of recipient site | 1, 4, 8 and 16 weeks post-operatively
Plasma bupivacaine levels | Before bolus and at 0.5, 1, 6, 12 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hayes JA, Forrest CR, Walsh W, Petroz GC, Adeli K, Bissonnette B. Continuous bupivacaine infusion post-iliac crest bone graft harvesting in pediatric cleft surgery: role and comparison with ketorolac. Cleft Palate Craniofac J. 2011 Sep;48(5):532-7. doi: 10.1597/10-148. Epub 2010 Nov 23. PMID 21091369